CLINICAL TRIAL: NCT01548417
Title: Medication Development in Alcoholism: Investigating Glucocorticoid Antagonists
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, PI, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: AA012602-11A1; 2R01AA012602-11A1 (NIH)
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Alcoholism
Keywords: Alcohol; Relapse
MeSH Terms: conditions — Alcoholism; Recurrence | interventions — Mifepristone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Korlym (mifepristone) (Active Comparator): 600 mg daily taken orally for one week
  Interventions: Drug: Korlym (mifepristone)
- Sugar Pill (Placebo Comparator): placebo pill daily taken orally for one week
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Korlym (mifepristone) — 600 mg/day, oral pill, 7 days
  Other Names: Mifepristone; C-1073; Mifeprex; RU-486
  Arms: Korlym (mifepristone)
Drug: Sugar Pill — 600 mg/day, oral pill, 7 days
  Other Names: Placebo
  Arms: Sugar Pill

SUMMARY:
The primary hypotheses under test are that alcohol dependent subjects treated with mifepristone will report decreased craving for alcohol following alcohol exposure in the laboratory and report significantly less drinking under naturalistic conditions, than those treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, 18-65 years of age
* Meets Diagnostic and Statistical Manual of Mental Disorders Fourth Addition (DSM-IV) criteria for current alcohol dependence
* Subjects will not be seeking treatment because the medication studies are not treatment trials
* Subjects must be abstinent a minimum of 3 days (but not more than 7 days) prior to the human lab session
* Negative Breath Alcohol Concentration (BAC) and a Clinical Institute Withdrawal Assessment-Alcohol (CIWA-A) score of < 8 at screening and time of lab session to eliminate acute alcohol or withdrawal effects on dependent measures
* Subjects must be able to complete and understand questionnaires and study procedures in English and sign an informed consent

Exclusion Criteria:

* Significant medical disorders that will increase potential risk or interfere with study participation as determined by the Study Physician
* Female subjects with childbearing potential who are pregnant, nursing, or refuse to use double barrier (non-hormonal) methods of birth control for the duration of the study and one month thereafter
* Meets DSM-IV criteria for a major Axis I disorder including mood or anxiety disorders or substance dependence disorders other than alcohol or nicotine dependence
* History of allergy or hypersensitivity to the study drugs or the ingredients
* Treatment within the month prior to screening with 1.) an investigational drug or vaccine; 2.) drugs that may influence study outcomes, e.g., disulfiram (Antabuse), naltrexone (ReVia), acamprosate (Campral), anticonvulsants, antidepressants.
* In need of or currently taking any psychoactive medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Mason, PhD, Principal Investigator — The Scripps Research Institute
Locations (1):
- The Scripps Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vendruscolo LF, Estey D, Goodell V, Macshane LG, Logrip ML, Schlosburg JE, McGinn MA, Zamora-Martinez ER, Belanoff JK, Hunt HJ, Sanna PP, George O, Koob GF, Edwards S, Mason BJ. Glucocorticoid receptor antagonism decreases alcohol seeking in alcohol-dependent individuals. J Clin Invest. 2015 Aug 3;125(8):3193-7. doi: 10.1172/JCI79828. Epub 2015 Jun 29. PMID 26121746
- See also: Laboratory Website Contact Form — http://alcoholismmarijuanatreatment.com/contact-us/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for study participation at the Laboratory of Clinical Psychopharmacology at The Scripps Research Institute in La Jolla, CA from 03/16/2012-03/14/2014. One Hundred twenty nine non-treatment seeking, paid volunteers signed informed consent, Fifty six subjects were enrolled, and Fifty four subjects completed the study.
Pre-assignment Details: Sixty six subjects were excluded from study participation due to exclusionary criteria, 2 subjects did not return after Visit 1, 4 subjects withdrew consent (2 for time constraints following Visit 1, 1 due to social motivations, 1 due to moving out of state), and 1 subject left the lab during Visit 1 when asked to provide a urine sample.
Groups:
- Sugar Pill: Sugar Pill: placebo, oral pill, 7 days
Period: Overall Study
Arm/Group | Korlym (Mifepristone) | Sugar Pill
Started | 28 | 28
Completed | 28 | 26
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Sugar Pill: placebo, oral pill, 7 days
- Total: Total of all reporting groups
Arm/Group | Korlym (Mifepristone) | Placebo | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (11.4) | 36.9 (11.2) | 39.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 23 | 20 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 23 | 21 | 44
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
DSM-V symptom count [Mean (Standard Deviation); unit: number of symptoms] — Diagnostic and Statistical Manual, 5th edition (DSM-V) requires 2 of 11 symptoms for a diagnosis of Alcohol Use Disorder.
  number of symptoms | 6.2 (2.3) | 6.9 (2.1) | 6.5 (2.2)
Years of heavy drinking [Mean (Standard Deviation); unit: years] | 15.0 (11) | 14.0 (8.9) | 14.5 (9.9)
DSM-IV symptom count [Mean (Standard Deviation); unit: number of symptoms] — Diagnostic and Statistical Manual, 4th edition (DSM-IV ) criteria for current Alcohol Dependence defined as three or more symptoms of dependence.
  number of symptoms | 4.7 (1.5) | 5.1 (1.5) | 4.8 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Craving to Drink
Description: Visual Analog Scale (VAS) scores of craving severity in response to in vivo alcohol cues. Higher scores indicate greater craving severity with a minimum score of 0 and a maximum score of 80.
Time Frame: 1 week
Population: 1 participant who completed the study had missing VAS scores.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Korlym (Mifepristone) | Sugar Pill
Number analyzed (Participants) | 27 | 26
units on a scale | 36.5 (1.5) | 42.9 (1.5)
Statistical Analysis 1: Comparison: Korlym (Mifepristone) vs Sugar Pill; Linear Mixed Effects Modeling (MEM) with Restricted Maximum Likelihood estimation was used to measure differences in alcohol-cued craving; Test type: Superiority or Other; p = .003, Mixed Models Analysis

2. Secondary Outcome: Drinking
Description: Number of standard drinks per week using the Timeline Followback Interview. Total number of alcoholic drinks consumed per week with a minimum value of 0 and a maximum value of 70.
Time Frame: 2 weeks
Population: Three randomized subjects who met exclusionary criteria were not included in the regression analysis for drinking: two subjects were excluded for unreliable reporting and one subject was excluded for being treatment seeking.
Measure: Mean (Standard Error); unit: alcoholic drinks per week
Arm/Group | Korlym (Mifepristone) | Sugar Pill
Number analyzed (Participants) | 26 | 25
alcoholic drinks per week | 27.661 (3.176) | 38.175 (3.239)
Statistical Analysis 1: Comparison: Korlym (Mifepristone) vs Sugar Pill; Linear Mixed Effect Modeling (MEM) with Restricted Maximum Likelihood estimation was used to measure differences in changes in drinking; Test type: Superiority or Other; p = .05, Mixed Models Analysis
Statistical Analysis 2: Comparison: Korlym (Mifepristone) vs Sugar Pill; Data represent the estimated marginal mean + or - SEM. *P<0.05, mifepristone vs. placebo (linear mixed effects modeling); Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at all five study visits, an average duration of 6 weeks.
Description: Adverse events, both serious and other, were documented at all five study visits by the Medical Assistant on the adverse events case report form.
Arm/Group | Korlym (Mifepristone) | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 12/28 | 8/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Korlym (Mifepristone) (N=28) | Sugar Pill (N=26)
Cold Symptoms (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dizzy/Foggy (Nervous system disorders) | 3 | 1
Abrasions/Bruises (Skin and subcutaneous tissue disorders) | 2 | 1
Muscle Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Fatigue (General disorders) | 3 | 1
Nausea/Gastrointestinal upset (Gastrointestinal disorders) | 3 | 1
Headache (General disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No